CLINICAL TRIAL: NCT00554164
Title: Positron Emission Tomography Guided Therapy of Aggressive Non-Hodgkin's Lymphomas
Acronym: PETAL
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Essen (Other)
Collaborators: Deutsche Krebshilfe e.V., Bonn (Germany) (Other)
Responsible Party: Principal Investigator, Ulrich Duehrsen, Prof. Dr. Ulrich Duehrsen, University Hospital, Essen
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PETAL trial; EudraCT-Number 2006-001641-33; Krebshilfe Grant 107592
Record Dates: First submitted 2007-11-05; First posted 2007-11-06 (Estimated); Last update posted 2017-05-05 (Actual); Status verified 2017-05

CONDITIONS: Lymphoma, High-grade
Keywords: Aggressive non-Hodgkin's lymphoma; Positron emission tomography; Chemotherapy
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — R-CHOP protocol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- B1 (Active Comparator): Six cycles of the (R-)CHOP regimen.
  Interventions: Drug: (R-)CHOP protocol
- B2 (Experimental): Six blocks of the B-ALL protocol.
  Interventions: Drug: B-ALL protocol
- A1 (Active Comparator): Four cycles of the (R-)CHOP regimen.
  Interventions: Drug: (R-)CHOP protocol
- A2 (Active Comparator): Four cycles of the (R-)CHOP regimen plus two additional doses rituximab.
  Interventions: Drug: (R-)CHOP protocol

INTERVENTIONS:
Drug: (R-)CHOP protocol — Patients with a persistently positive interim-PET scan assigned to arm B1 will receive another six cycles of the (R-)CHOP regimen (rituximab, cyclophosphamide, doxorubicine, vincristine, prednisone).
  Arms: B1
Drug: B-ALL protocol — Patients with a persistently positive interim-PET scan assigned to arm B2 will receive six blocks of the B-ALL protocol (rituximab, methotrexate, ifosfamide, etoposide, cytarabine, vincristine, cyclophosphamide, doxorubicine, vindesine, dexamethasone).
  Arms: B2
Drug: (R-)CHOP protocol — Patients with a negative interim-PET scan assigned to arm A1 will receive another four cycles of the (R-)CHOP regimen (rituximab, cyclophosphamide, doxorubicine, vincristine, prednisone). Arm A1 was closed when the number of patients required for the randomisation between arms A1 and A2 was reached.
  Arms: A1
Drug: (R-)CHOP protocol — Patients with a negative interim-PET scan assigned to arm A2 will receive another four cycles of the (R-)CHOP regimen (rituximab, cyclophosphamide, doxorubicine, vincristine, prednisone) plus two additional doses rituximab. Since the number of patients required for the randomisation between arms A1 and A2 has been reached, all patients with a negative interim-PET scan are treated according to arm A2.
  Arms: A2

SUMMARY:
The main purpose of the PETAL trial is to determine whether patients with aggressive non-Hodgkin's lymphomas with a persistently positive PET scan after two cycles of chemotherapy benefit from a change of the treatment protocol.

DETAILED DESCRIPTION:
Positron emission tomography performed after two cycles of (R-)CHOP chemotherapy (interim-PET) has been shown to predict long-term outcome in patients with aggressive non-Hodgkin's lymphomas. Patients with early normalization of pathological PET findings have an excellent prognosis, while patients with a persistently pathological PET scan have a high risk of non-response or relapse.

Patients with a negative interim-PET scan (part A of the trial) will be randomized to receive either another four cycles of the (R-)CHOP regimen (arm A1) or four cycles of the (R-)CHOP regimen plus two additional doses of rituximab (arm A2). Randomisation in part A of the trial was stopped when the number of patients required was reached (128 patients in each treatment arm). Since then patients have been uniformly treated according to arm A2.

Patients with a persistently positive interim-PET scan (part B of the trial) will be randomized to either continue treatment with another six (R-)CHOP cycles (arm B1) or switch to an alternative protocol used for the treatment of Burkitt's lymphoma (arm B2: six blocks according to the so-called B-ALL protocol of the German ALL study group).

Patients refractory to or relapsing within two years after treatment according to parts A or B of the trial will receive age-adapted salvage protocols (patients < 60 years: high-dose chemotherapy with autologous stem cell transplantation; patients > 60 years: (R-)ESHAP protocol)(part C of the trial).

ELIGIBILITY:
Inclusion Criteria:

* Aggressive B-cell or T-cell non-Hodgkin's lymphoma
* Pathological pre-treatment PET scan
* Performance status ECOG 0-3
* Age 18 - 80 years
* Ability to understand the purpose of the study and act accordingly
* Willingness to use adequate contraception
* Informed consent

Exclusion Criteria:

* Burkitt's lymphoma
* Primary central nervous system lymphoma
* Previous chemo- and/or radiotherapy
* Other cancer within preceding 5 years
* HIV infection, active viral hepatitis or other uncontrolled infection
* Other medical conditions precluding administration of planned therapy
* Pregnancy or lactation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1073 (Actual)
Dates: Start 2007-11; Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Time to treatment failure | Two years

SECONDARY OUTCOMES:
Response rate, overall survival, disease-free survival, toxicity, quality of life | Two years

CONTACTS AND LOCATIONS:
Overall Officials: Ulrich Duehrsen, Prof. Dr., Principal Investigator — Department of Hematology, University Hospital Essen, Hufelandstrasse 55, 45122 Essen, Germany
Locations (1):
- Department of Hematology, University Hospital Essen, Essen, Germany

REFERENCES:
- [Derived] Duhrsen U, Bockisch A, Hertenstein B, Karsten IE, Kroschinsky F, Heuser M, Hochhaus A, Hoffkes HG, Behringer D, Prange-Krex G, Tometten M, Grieshammer M, Grigoleit GU, Schmalz O, Jordan K, Bernhard H, Gaska T, Giagounidis A, Schroers R, Martens UM, Held G, Klapper W, Jockel KH, Nonnemacher M, Huttmann A; PETAL Trial Investigators. Response-guided first-line therapy and treatment of relapse in aggressive lymphoma: 10-year follow-up of the PETAL trial. Blood Neoplasia. 2024 May 21;1(3):100018. doi: 10.1016/j.bneo.2024.100018. eCollection 2024 Sep. PMID 40453056
- [Derived] Duhrsen U, Prange-Krex G, Moeller R, Held H, Heil G, Schwarzer A, Mahlmann S, Dienst A, Sandmann M, Maschmeyer G, Schutte J, Hahn D, Heike M, Nonnemacher M, Hanoun C, Huttmann A; PETAL trial investigators. Health-related quality of life in patients with aggressive non-Hodgkin lymphoma: results from the PETAL trial. Ann Hematol. 2025 May;104(5):2831-2845. doi: 10.1007/s00277-025-06402-1. Epub 2025 May 21. PMID 40397196
- [Derived] Broecker-Preuss M, Becher-Boveleth N, Muller SP, Huttmann A, Hanoun C, Grafe H, Richter J, Klapper W, Rekowski J, Bockisch A, Duhrsen U. Impact of germline polymorphisms in genes regulating glucose uptake on positron emission tomography findings and outcome in diffuse large B-cell lymphoma: results from the PETAL trial. J Cancer Res Clin Oncol. 2022 Oct;148(10):2611-2621. doi: 10.1007/s00432-021-03796-z. Epub 2021 Oct 27. PMID 34708297
- [Derived] Kaddu-Mulindwa D, Altmann B, Held G, Angel S, Stilgenbauer S, Thurner L, Bewarder M, Schwier M, Pfreundschuh M, Loffler M, Menhart K, Grosse J, Ziepert M, Herrmann K, Duhrsen U, Huttmann A, Barbato F, Poeschel V, Hellwig D. FDG PET/CT to detect bone marrow involvement in the initial staging of patients with aggressive non-Hodgkin lymphoma: results from the prospective, multicenter PETAL and OPTIMAL>60 trials. Eur J Nucl Med Mol Imaging. 2021 Oct;48(11):3550-3559. doi: 10.1007/s00259-021-05348-6. Epub 2021 Apr 29. PMID 33928400
- [Derived] Schmitz C, Rekowski J, Reinke S, Muller SP, Huttmann A, Klapper W, Duhrsen U. Metabolic tumor volume, cancer cell fraction, and prognosis - the case of T-cell/histiocyte-rich large B-cell lymphoma. Leuk Lymphoma. 2020 Jun;61(6):1372-1379. doi: 10.1080/10428194.2020.1713319. Epub 2020 Feb 5. PMID 32022621
- [Derived] Schmitz C, Huttmann A, Muller SP, Hanoun M, Boellaard R, Brinkmann M, Jockel KH, Duhrsen U, Rekowski J. Dynamic risk assessment based on positron emission tomography scanning in diffuse large B-cell lymphoma: Post-hoc analysis from the PETAL trial. Eur J Cancer. 2020 Jan;124:25-36. doi: 10.1016/j.ejca.2019.09.027. Epub 2019 Nov 9. PMID 31710995
- [Derived] Kurtz DM, Scherer F, Jin MC, Soo J, Craig AFM, Esfahani MS, Chabon JJ, Stehr H, Liu CL, Tibshirani R, Maeda LS, Gupta NK, Khodadoust MS, Advani RH, Levy R, Newman AM, Duhrsen U, Huttmann A, Meignan M, Casasnovas RO, Westin JR, Roschewski M, Wilson WH, Gaidano G, Rossi D, Diehn M, Alizadeh AA. Circulating Tumor DNA Measurements As Early Outcome Predictors in Diffuse Large B-Cell Lymphoma. J Clin Oncol. 2018 Oct 1;36(28):2845-2853. doi: 10.1200/JCO.2018.78.5246. Epub 2018 Aug 20. PMID 30125215
- [Derived] Duhrsen U, Muller S, Hertenstein B, Thomssen H, Kotzerke J, Mesters R, Berdel WE, Franzius C, Kroschinsky F, Weckesser M, Kofahl-Krause D, Bengel FM, Durig J, Matschke J, Schmitz C, Poppel T, Ose C, Brinkmann M, La Rosee P, Freesmeyer M, Hertel A, Hoffkes HG, Behringer D, Prange-Krex G, Wilop S, Krohn T, Holzinger J, Griesshammer M, Giagounidis A, Raghavachar A, Maschmeyer G, Brink I, Bernhard H, Haberkorn U, Gaska T, Kurch L, van Assema DME, Klapper W, Hoelzer D, Geworski L, Jockel KH, Scherag A, Bockisch A, Rekowski J, Huttmann A; PETAL Trial Investigators. Positron Emission Tomography-Guided Therapy of Aggressive Non-Hodgkin Lymphomas (PETAL): A Multicenter, Randomized Phase III Trial. J Clin Oncol. 2018 Jul 10;36(20):2024-2034. doi: 10.1200/JCO.2017.76.8093. Epub 2018 May 11. PMID 29750632
- [Derived] Huttmann A, Muller S, Jockel KH, Duhrsen U. Pitfalls of interim positron emission tomography scanning in diffuse large B-cell lymphoma. J Clin Oncol. 2010 Sep 20;28(27):e488-9; author reply e490-1. doi: 10.1200/JCO.2010.29.5428. Epub 2010 Jul 19. No abstract available. PMID 20644097
- [Derived] Duhrsen U, Huttmann A, Jockel KH, Muller S. Positron emission tomography guided therapy of aggressive non-Hodgkin lymphomas--the PETAL trial. Leuk Lymphoma. 2009 Nov;50(11):1757-60. doi: 10.3109/10428190903308031. PMID 19863177